CLINICAL TRIAL: NCT00000653
Title: A Trial of Two Doses of 2',3'-Dideoxycytidine (ddC) in the Treatment of Children With Symptomatic HIV Infection Who Are Intolerant of AZT and/or Who Show Progressive Disease While on AZT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 138; 11113 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zalcitabine

INTERVENTIONS:
Drug: Zalcitabine

SUMMARY:
To evaluate and compare the long-term (48-177 weeks) safety, tolerance, and efficacy of two doses of zalcitabine ( dideoxycytidine; ddC ) taken orally every 8 hours in children with symptomatic HIV infection who have one of the following: intolerance to zidovudine ( AZT ) (development of toxicity during prolonged AZT therapy), demonstrated disease progression after 6 months of AZT therapy, OR both AZT intolerance and disease progression after 6 months of AZT therapy.

As useful as AZT appears to be in the treatment of patients infected with HIV, it is associated with significant toxicity in some patients, and it does not prevent ultimate progression to AIDS and eventual mortality. Thus, there is a clear need for new antiretroviral drugs, and ddC is one such promising agent.

DETAILED DESCRIPTION:
As useful as AZT appears to be in the treatment of patients infected with HIV, it is associated with significant toxicity in some patients, and it does not prevent ultimate progression to AIDS and eventual mortality. Thus, there is a clear need for new antiretroviral drugs, and ddC is one such promising agent.

Patients receive oral ddC for 48 to 177 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Procrit.
* Amphotericin B (1 mg/kg up to 5 days/week).
* Prophylaxis treatment as per ACTG recommendations for Pneumocystis carinii pneumonia.
* Acyclovir (up to 1000 mg/day PO; for > 1000 mg/day PO or for any IV dose, suggest interrupting ddC).
* Ketoconazole (up to 10 mg/kg/day).
* Nystatin.
* Aspirin, acetaminophen, sedatives, and barbiturates (for up to 72 hours).
* Isoniazid (INH), if there is no evidence of peripheral neuropathy at entry. Children should receive pyridoxine, 25
* 50 mg/day to avoid possible INH-associated neuropathy.
* Trimethoprim / sulfamethoxazole (T/S).
* Immunoglobulin therapy.
* Aerosolized pentamidine.
* Drugs with little nephro-, hepato-, cytotoxicity that the patient has been taking and tolerating well for an ongoing condition.

Concurrent Treatment:

Allowed:

* Immunoglobulin therapy.
* Nutritional support (for children with wasting syndrome and/or malnutritional) including hyperalimentation (TPN) of dietary supplements.

AMENDED:

* Patients enrolled in ACTG 051 may participate in ACTG 138 if they show intolerance to AZT or show disease progression after 6 months of AZT therapy and meet entry criteria for the study.

ORIGINAL design:

* Patients enrolled in ACTG protocols 051 or 128 must meet study end points or meet protocol definitions for being permanently off zidovudine (AZT) before enrolling in this protocol.

Patients must have the following:

* Absence of acute opportunistic infection at time of entry.
* However, if patient is successfully treated for opportunistic infection and has remained stable for 2 weeks after treatment, the patient is then allowed to enter the study. Children receiving maintenance therapy for > 4 weeks are eligible.
* Parent or guardian available to give written informed consent.

Allowed at time of study entry:

* Prophylaxis treatment as per ACTG recommendations, for Pneumocystis carinii pneumonia (PCP).
* Immunoglobulin therapy.

Prior Medication:

AMENDED:

* AZT or ddI up until study entry, other antiretrovirals up until 4 weeks of study entry

Allowed:

* Zidovudine (AZT) within 4 weeks of entry.
* Dideoxyinosine (ddI) within 43 weeks of entry if no peripheral neuropathy has been observed while receiving ddI.
* Other toxicities observed while on ddI must resolve to level 2 or better before patient can begin treatment with ddC.
* Vitamin, folate, iron supplements.

Exclusion Criteria

Co-existing Condition:

AMENDED:

* 04-25-91 Additional excluded symptoms and conditions:
* Symptomatic cardiomyopathy.
* Seizures which are not well controlled by ongoing anticonvulsant therapy.
* Active malignancy requiring concomitant chemotherapy.
* Symptomatic pancreatitis.
* Grade I or greater peripheral neuropathy.
* Receiving concomitant zidovudine (AZT).
* Patients with the following conditions or symptoms are excluded:
* Acute bacterial infections requiring IV or oral antibiotic treatment at time of entry.
* Known hypersensitivity to dideoxycytidine (ddC).

Concurrent Medication:

Excluded:

* Other antiviral agents, biological modifiers, and investigational medications.
* Drugs with potential to cause peripheral neuropathy, including chloramphenicol, iodoquinol, phenytoin, ethionamide, gold, ribavirin, vincristine, cisplatin, dapsone, disulfiram, glutethimide, hydralazine, metronidazole, nitrofurantoin.

Patients with the following are excluded:

* Acute bacterial infections requiring IV or oral antibiotic treatment at time of entry.
* Known hypersensitivity to dideoxycytidine (ddC).
* Active opportunistic infection requiring treatment with an excluded concomitant medication.

Prior Medication:

Excluded:

* Antiretroviral agents (other than zidovudine (AZT) or didanosine (ddI)) within 4 weeks of entry.
* Immunomodulating agents such as interferons, isoprinosine, or interleukin-2 within 2 weeks of entry.
* Any other experimental therapy, drugs that cause prolonged neutropenia, significant nephrotoxicity, or peripheral neuropathy within 1 week of entry.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140
Dates: Study Completion 1995-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spector SA, Study Chair
Locations (35):
- United States (32):
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Emory Univ. School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Atlanta, Georgia
  - Cook County Hosp., Chicago, Illinois
  - Univ. of Illinois College of Medicine at Chicago, Dept. of Peds., Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - UMDNJ - Robert Wood Johnson, New Brunswick, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - North Shore-Long Island Jewish Health System, Dept. of Peds., Great Neck, New York
  - Schneider Children's Hosp., Div. of Infectious Diseases, New Hyde Park, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - UNC at Chapel Hill School of Medicine - Dept. of Peds., Div. of Immunology & Infectious Diseases, Chapel Hill, North Carolina
  - DUMC Ped. CRS, Durham, North Carolina
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - Texas Children's Hosp. CRS, Houston, Texas
- Puerto Rico (3):
  - Univ. Hosp. Ramón Ruiz Arnau, Dept. of Peds., Bayamón
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891
- [Background] Spector SA, Blanchard S, Connor EM, Salgo MP, McNamara J. Results of a clinical trial comparing two doses of 2'3'-dideoxycytidine (ddC) in the treatment of children with symptomatic human immunodeficiency virus (HIV) infection who were intolerant or had failed zidovudine (ZDV) therapy (ACTG 138). The Pediatric AIDS Clinical Trials Group. American Pediatric Society 104th annual meeting and Society for Pediatric Research 63rd annual meeting; 1994 May 2-5; Seattle. Pediatr AIDS HIV Infect. 1994 Oct;5(5):323 (unnumbered abstract)